CLINICAL TRIAL: NCT03768089
Title: A Phase 1/2 Study of VX-121 in Healthy Subjects and in Subjects With Cystic Fibrosis
Brief Title: Study of VX-121 in Healthy Subjects and in Subjects With Cystic Fibrosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX17-121-001; 2018-000126-55 (EudraCT Number)
Record Dates: First submitted 2018-12-05; First posted 2018-12-07 (Actual); Results first posted 2022-07-14 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-06

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Suspensions; tezacaftor, ivacaftor drug combination; ivacaftor; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (18):
- Part A: Pooled Placebo (Cohorts A1-5; Except A3) (Placebo Comparator): Participants received single dose of placebo matched to VX-121.
  Interventions: Drug: Placebo (matched to VX-121 suspension)
- Part A: VX-121 (Cohort A1) (Experimental): Participants received single dose of VX-121 10 milligrams (mg).
  Interventions: Drug: VX-121 (Suspension)
- Part A: VX-121 (Cohort A2) (Experimental): Participants received single dose of VX-121 20 mg.
  Interventions: Drug: VX-121 (Suspension)
- Part A: VX-121 (Cohort A3) (Experimental): Participants received single dose of VX-121 5 mg or matched placebo without milk, followed by open label VX-121 5 mg with milk.
  Interventions: Drug: Placebo (matched to VX-121 suspension); Drug: VX-121 (Suspension)
- Part A: VX-121 (Cohort A4) (Experimental): Participants received single dose of VX-121 40 mg.
  Interventions: Drug: VX-121 (Suspension)
- Part A: VX-121 (Cohort A5) (Experimental): Participants received single dose of VX-121 60 mg.
  Interventions: Drug: VX-121 (Suspension)
- Part A: VX-121 (Cohort A9) (Experimental): Participants received single dose of VX-121 10 mg suspension on Day 1, VX-121 10 mg tablet on Day 9, followed by VX-121 10 mg tablet with milk on Day 17.
  Interventions: Drug: VX-121 (Suspension); Drug: VX-121 (Tablet)
- Part B: Pooled Placebo (Cohorts B1-4) (Placebo Comparator): Participants received placebo matched to VX-121 for 10 days.
  Interventions: Drug: Placebo (matched to VX-121 suspension)
- Part B: VX-121 (Cohort B1) (Experimental): Participants received VX-121 10 mg once daily (qd) for 10 days.
  Interventions: Drug: VX-121 (Suspension)
- Part B: VX-121 (Cohort B2) (Experimental): Participants received VX-121 20 mg qd for 10 days.
  Interventions: Drug: VX-121 (Suspension)
- Part B: VX-121 (Cohort B3) (Experimental): Participants received VX-121 40 mg qd for 10 days.
  Interventions: Drug: VX-121 (Suspension)
- Part B: VX-121 (Cohort B4) (Experimental): Participants received VX-121 60 mg qd for 10 days.
  Interventions: Drug: VX-121 (Suspension)
- Part C: Pooled Placebo (Cohorts C1-3) (Placebo Comparator): Participants received placebo matched to VX-121/TEZ/IVA for 14 days.
  Interventions: Drug: Placebo (matched to VX-121 suspension); Drug: Placebo (matched to TEZ/IVA); Drug: Placebo (matched to IVA)
- Part C: VX-121 (Cohort C1) (Experimental): Participants received VX-121 10 mg qd/TEZ 100 mg qd/IVA 150 mg every 12 hours (q12h) for 14 days.
  Interventions: Drug: VX-121 (Suspension); Drug: TEZ/IVA; Drug: IVA
- Part C: VX-121 (Cohort C2) (Experimental): Participants received VX-121 20 mg qd/TEZ 100 mg qd/IVA 150 mg q12h for 14 days.
  Interventions: Drug: VX-121 (Suspension); Drug: TEZ/IVA; Drug: IVA
- Part C: VX-121 (Cohort C3) (Experimental): Participants received VX-121 5 mg qd/TEZ 100 mg qd/IVA 150 mg q12h for 14 days.
  Interventions: Drug: VX-121 (Suspension); Drug: TEZ/IVA; Drug: IVA
- Part D: Placebo (Placebo Comparator): Participants received placebo matched to VX-121/TEZ/IVA for 4 weeks.
  Interventions: Drug: Placebo (matched to TEZ/IVA); Drug: Placebo (matched to IVA); Drug: Placebo (matched to VX-121 tablet)
- Part D: VX-121/TEZ/IVA (Experimental): Participants received VX-121 5 mg qd/TEZ 100 mg qd/IVA 150 mg q12h for 4 weeks.
  Interventions: Drug: TEZ/IVA; Drug: IVA; Drug: VX-121 (Tablet)

INTERVENTIONS:
Drug: Placebo (matched to VX-121 suspension) — Placebo matched to VX-121 suspension for oral administration.
  Arms: Part A: Pooled Placebo (Cohorts A1-5; Except A3); Part A: VX-121 (Cohort A3); Part B: Pooled Placebo (Cohorts B1-4); Part C: Pooled Placebo (Cohorts C1-3)
Drug: VX-121 (Suspension) — Suspension for oral administration.
  Arms: Part A: VX-121 (Cohort A1); Part A: VX-121 (Cohort A2); Part A: VX-121 (Cohort A3); Part A: VX-121 (Cohort A4); Part A: VX-121 (Cohort A5); Part A: VX-121 (Cohort A9); Part B: VX-121 (Cohort B1); Part B: VX-121 (Cohort B2); Part B: VX-121 (Cohort B3); Part B: VX-121 (Cohort B4); Part C: VX-121 (Cohort C1); Part C: VX-121 (Cohort C2); Part C: VX-121 (Cohort C3)
Drug: TEZ/IVA — Fixed-dose combination tablet for oral administration.
  Other Names: VX-661/VX-770; tezacaftor/ivacaftor
  Arms: Part C: VX-121 (Cohort C1); Part C: VX-121 (Cohort C2); Part C: VX-121 (Cohort C3); Part D: VX-121/TEZ/IVA
Drug: IVA — Tablet for oral administration.
  Other Names: VX-770; ivacaftor
  Arms: Part C: VX-121 (Cohort C1); Part C: VX-121 (Cohort C2); Part C: VX-121 (Cohort C3); Part D: VX-121/TEZ/IVA
Drug: Placebo (matched to TEZ/IVA) — Placebo matched to TEZ/IVA for oral administration.
  Arms: Part C: Pooled Placebo (Cohorts C1-3); Part D: Placebo
Drug: Placebo (matched to IVA) — Placebo matched to IVA for oral administration.
  Arms: Part C: Pooled Placebo (Cohorts C1-3); Part D: Placebo
Drug: VX-121 (Tablet) — Tablet for oral administration.
  Arms: Part A: VX-121 (Cohort A9); Part D: VX-121/TEZ/IVA
Drug: Placebo (matched to VX-121 tablet) — Placebo matched to VX-121 tablet for oral administration.
  Arms: Part D: Placebo

SUMMARY:
The purpose of this study is to evaluate safety and tolerability of VX-121 in healthy subjects and in subjects with cystic fibrosis (CF).

ELIGIBILITY:
Key Inclusion Criteria:

* Part A, B, and C: Healthy Volunteers

  * Female subjects must be of non-childbearing potential
  * Between the ages of 18 and 55 years, inclusive
  * Body mass index (BMI) of 18.0 to 32.0 kg/m2, inclusive, and a total body weight >50 kg
* Part D: Subjects with CF

  * Heterozygous for F508del and an MF mutation (F/MF)
  * FEV1 value ≥40% and ≤90% of predicted mean for age, sex, and height
  * Body weight ≥35 kg

Key Exclusion Criteria:

* Part A, B and C: Healthy Volunteers

  * Any condition possibly affecting drug absorption
  * History of febrile illness or other acute illness within 5 days before the first study drug dose
* Part D: Subjects with CF

  * History of clinically significant cirrhosis with or without portal hypertension
  * History of solid organ or hematological transplantation
  * Lung infection with organisms associated with a more rapid decline in pulmonary status

Other protocol defined Inclusion/Exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2019-05-03 (Actual); Study Completion 2019-05-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- Netherlands (5):
  - Academic Medical Center, Amsterdam
  - PRA Health Sciences Onderzoekscentrum UMCG, Groningen
  - UMC St. Radboud, Nijmegen
  - Erasmus Medical Center, Rotterdam
  - HagaZiekenhuis van den Haag, The Hague
- United Kingdom (2):
  - Heart of England NHS Foundation Trust, Birmingham Heartlands Hospital, Birmingham
  - The Medicines Evaluation Unit, Manchester

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 115 unique participants enrolled in this study.
Pre-assignment Details: This study included 4 parts: Parts A, B, and C were conducted in healthy adult participants; Part D was conducted in adult cystic fibrosis (CF) participants.
Period: Part A
Arm/Group | Part A: Pooled Placebo (Cohorts A1-5; Except A3) | Part A: VX-121 (Cohort A1) | Part A: VX-121 (Cohort A2) | Part A: VX-121 (Cohort A3) | Part A: VX-121 (Cohort A4) | Part A: VX-121 (Cohort A5) | Part A: VX-121 (Cohort A9) | Part B: Pooled Placebo (Cohorts B1-4) | Part B: VX-121 (Cohort B1) | Part B: VX-121 (Cohort B2) | Part B: VX-121 (Cohort B3) | Part B: VX-121 (Cohort B4) | Part C: Pooled Placebo (Cohorts C1-3) | Part C: VX-121 (Cohort C1) | Part C: VX-121 (Cohort C2) | Part C: VX-121 (Cohort C3) | Part D: Placebo | Part D: VX-121/TEZ/IVA
Started | 8 | 5 | 6 | 6 | 6 | 6 | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Safety Set (Received at least 1 dose of study drug.) | 8 | 5 | 6 | 6 | 6 | 6 | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 8 | 5 | 6 | 6 | 5 | 6 | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part B
Arm/Group | Part A: Pooled Placebo (Cohorts A1-5; Except A3) | Part A: VX-121 (Cohort A1) | Part A: VX-121 (Cohort A2) | Part A: VX-121 (Cohort A3) | Part A: VX-121 (Cohort A4) | Part A: VX-121 (Cohort A5) | Part A: VX-121 (Cohort A9) | Part B: Pooled Placebo (Cohorts B1-4) | Part B: VX-121 (Cohort B1) | Part B: VX-121 (Cohort B2) | Part B: VX-121 (Cohort B3) | Part B: VX-121 (Cohort B4) | Part C: Pooled Placebo (Cohorts C1-3) | Part C: VX-121 (Cohort C1) | Part C: VX-121 (Cohort C2) | Part C: VX-121 (Cohort C3) | Part D: Placebo | Part D: VX-121/TEZ/IVA
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 6 | 6 | 6 (One participant who participated in A2 also participated in B3.) | 6 | 0 | 0 | 0 | 0 | 0 | 0
Safety Set (Received at least 1 dose of study drug.) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 6 | 6 | 6 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 6 | 6 | 6 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part C
Arm/Group | Part A: Pooled Placebo (Cohorts A1-5; Except A3) | Part A: VX-121 (Cohort A1) | Part A: VX-121 (Cohort A2) | Part A: VX-121 (Cohort A3) | Part A: VX-121 (Cohort A4) | Part A: VX-121 (Cohort A5) | Part A: VX-121 (Cohort A9) | Part B: Pooled Placebo (Cohorts B1-4) | Part B: VX-121 (Cohort B1) | Part B: VX-121 (Cohort B2) | Part B: VX-121 (Cohort B3) | Part B: VX-121 (Cohort B4) | Part C: Pooled Placebo (Cohorts C1-3) | Part C: VX-121 (Cohort C1) | Part C: VX-121 (Cohort C2) | Part C: VX-121 (Cohort C3) | Part D: Placebo | Part D: VX-121/TEZ/IVA
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 8 | 6 | 0 | 0
Safety Set (Received at least 1 dose of study drug.) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 7 | 6 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 7 | 6 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Randomized, Never Dosed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Period: Part D
Arm/Group | Part A: Pooled Placebo (Cohorts A1-5; Except A3) | Part A: VX-121 (Cohort A1) | Part A: VX-121 (Cohort A2) | Part A: VX-121 (Cohort A3) | Part A: VX-121 (Cohort A4) | Part A: VX-121 (Cohort A5) | Part A: VX-121 (Cohort A9) | Part B: Pooled Placebo (Cohorts B1-4) | Part B: VX-121 (Cohort B1) | Part B: VX-121 (Cohort B2) | Part B: VX-121 (Cohort B3) | Part B: VX-121 (Cohort B4) | Part C: Pooled Placebo (Cohorts C1-3) | Part C: VX-121 (Cohort C1) | Part C: VX-121 (Cohort C2) | Part C: VX-121 (Cohort C3) | Part D: Placebo | Part D: VX-121/TEZ/IVA
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 9
Safety Set (Received at least 1 dose of study drug.) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 9
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 9
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis population included all participants who received at least 1 dose of study drug. The participant who participated in Parts A2 and B3 counted only once in Part A: VX-121 (Cohort A2) reporting arm.
Groups:
- Part A: VX-121 (Cohort A1): Participants received single dose of VX-121 10 mg.
- Part A: Cohort A9: Participants received single dose of VX-121 10 mg suspension on Day 1, VX-121 10 mg tablet on Day 9, followed by VX-121 10 mg tablet with milk on Day 17.
- Part B: VX-121 (Cohort B1): Participants received VX-121 10 mg qd for 10 days.
- Part C: Pooled Placebo (Cohorts C1-3): Participants received placebo matched to VX-121/TEZ/IVA in for 14 days.
- Part C: VX-121 (Cohort C1): Participants received VX-121 10 mg qd/TEZ 100 mg qd/IVA 150 mg q12h for 14 days.
- Total: Total of all reporting groups
Arm/Group | Part A: Pooled Placebo (Cohorts A1-5; Except A3) | Part A: VX-121 (Cohort A1) | Part A: VX-121 (Cohort A2) | Part A: VX-121 (Cohort A3) | Part A: VX-121 (Cohort A4) | Part A: VX-121 (Cohort A5) | Part A: Cohort A9 | Part B: Pooled Placebo (Cohorts B1-4) | Part B: VX-121 (Cohort B1) | Part B: VX-121 (Cohort B2) | Part B: VX-121 (Cohort B3) | Part B: VX-121 (Cohort B4) | Part C: Pooled Placebo (Cohorts C1-3) | Part C: VX-121 (Cohort C1) | Part C: VX-121 (Cohort C2) | Part C: VX-121 (Cohort C3) | Part D: Placebo | Part D: VX-121/TEZ/IVA | Total
Number analyzed (Participants) | 8 | 5 | 6 | 6 | 6 | 6 | 8 | 9 | 6 | 6 | 5 | 6 | 6 | 6 | 7 | 6 | 3 | 9 | 114
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 5 | 6 | 6 | 6 | 6 | 8 | 9 | 6 | 6 | 5 | 6 | 6 | 6 | 7 | 6 | 3 | 9 | 114
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 5
  Male | 8 | 5 | 6 | 6 | 5 | 5 | 8 | 8 | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 3 | 8 | 109
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 5
  Not Hispanic or Latino | 8 | 5 | 5 | 5 | 6 | 5 | 7 | 9 | 6 | 6 | 5 | 6 | 6 | 5 | 7 | 6 | 3 | 9 | 109
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Asian | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 8
  White | 5 | 5 | 6 | 4 | 4 | 5 | 4 | 6 | 5 | 6 | 5 | 5 | 4 | 5 | 5 | 5 | 3 | 8 | 90
  More than one race | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 7
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability as Assessed by Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Time Frame: From Day 1 Through Safety Follow-up (up to Day 15 for Part A [except Cohorts A3 and A9], up to Day 26 for Cohort A3, up to Day 34 for Cohort A9, up to Day 20 for Part B, up to Day 24 for Part C and up to Week 9 for Part D)
Population: Safety Set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Part A: Pooled Placebo (Cohorts A1-5; Except A3) | Part A: VX-121 (Cohort A1) | Part A: VX-121 (Cohort A2) | Part A: VX-121 (Cohort A3) | Part A: VX-121 (Cohort A4) | Part A: VX-121 (Cohort A5) | Part A: VX-121 (Cohort A9) | Part B: Pooled Placebo (Cohorts B1-4) | Part B: VX-121 (Cohort B1) | Part B: VX-121 (Cohort B2) | Part B: VX-121 (Cohort B3) | Part B: VX-121 (Cohort B4) | Part C: Pooled Placebo (Cohorts C1-3) | Part C: VX-121 (Cohort C1) | Part C: VX-121 (Cohort C2) | Part C: VX-121 (Cohort C3) | Part D: Placebo | Part D: VX-121/TEZ/IVA
Number analyzed (Participants) | 8 | 5 | 6 | 6 | 6 | 6 | 9 | 9 | 6 | 6 | 6 | 6 | 6 | 6 | 7 | 6 | 3 | 9
participants
  Participants With TEAEs | 1 | 4 | 2 | 4 | 1 | 2 | 7 | 7 | 3 | 5 | 4 | 5 | 4 | 3 | 6 | 3 | 2 | 7
  Participants With SAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

2. Secondary Outcome: Part A: Maximum Observed Concentration (Cmax) of VX-121
Time Frame: Cohorts A1-5 (Except A3): Pre-dose up to 240 hours post-dose; Cohorts A3 and A9: Pre-dose up to 168 hours post-dose
Population: The pharmacokinetic (PK) set included all participants who received at least 1 dose of study drug and for whom the primary PK data are considered sufficient and interpretable.
Measure: Mean (Standard Deviation); unit: microgram per milliliter (mcg/mL)
Groups:
- Part A: VX-121 (Cohort A3: Without Milk): Participants received single dose of VX-121 5 mg without milk.
- Part A: VX-121 (Cohort A3: With Milk): Participants received single dose of VX-121 5 mg with milk.
- Part A: VX-121 (Cohort A9: Suspension): Participants received single dose of VX-121 10 mg suspension on Day 1.
- Part A: VX-121 (Cohort A9: Tablet Without Milk): Participants received single dose of VX-121 10 mg tablet without milk on Day 9.
- Part A: VX-121 (Cohort A9: Tablet With Milk): Participants received single dose of VX-121 10 mg tablet with milk on Day 17.
Arm/Group | Part A: VX-121 (Cohort A1) | Part A: VX-121 (Cohort A2) | Part A: VX-121 (Cohort A3: Without Milk) | Part A: VX-121 (Cohort A3: With Milk) | Part A: VX-121 (Cohort A4) | Part A: VX-121 (Cohort A5) | Part A: VX-121 (Cohort A9: Suspension) | Part A: VX-121 (Cohort A9: Tablet Without Milk) | Part A: VX-121 (Cohort A9: Tablet With Milk)
Number analyzed (Participants) | 5 | 6 | 5 | 5 | 6 | 6 | 8 | 8 | 8
microgram per milliliter (mcg/mL) | 0.134 (0.0295) | 0.247 (0.0515) | 0.0705 (0.0152) | 0.061 (0.0143) | 0.893 (0.216) | 1.04 (0.263) | 0.181 (0.0458) | 0.178 (0.0447) | 0.156 (0.0352)

3. Secondary Outcome: Part A: Area Under the Concentration Versus Time Curve From the Time of Dosing to the Last Measurable Concentration (AUC[0-last]) of VX-121
Time Frame: Cohorts A1-5 (Except A3): Pre-dose up to 240 hours post-dose; Cohorts A3 and A9: Pre-dose up to 168 hours post-dose
Population: PK set.
Measure: Mean (Standard Deviation); unit: microgram*hour per milliliter (mcg*h/mL)
Arm/Group | Part A: VX-121 (Cohort A1) | Part A: VX-121 (Cohort A2) | Part A: VX-121 (Cohort A3: Without Milk) | Part A: VX-121 (Cohort A3: With Milk) | Part A: VX-121 (Cohort A4) | Part A: VX-121 (Cohort A5) | Part A: VX-121 (Cohort A9: Suspension) | Part A: VX-121 (Cohort A9: Tablet Without Milk) | Part A: VX-121 (Cohort A9: Tablet With Milk)
Number analyzed (Participants) | 5 | 6 | 5 | 5 | 6 | 6 | 8 | 8 | 8
microgram*hour per milliliter (mcg*h/mL) | 7.72 (1.93) | 20.7 (7.03) | 6.32 (2.54) | 5.36 (2.09) | 72.2 (28.9) | 66.6 (9.18) | 15.7 (3.88) | 14.6 (3.85) | 13.1 (2.56)

4. Secondary Outcome: Part B: Maximum Observed Concentration (Cmax) of VX-121
Time Frame: Day 1, Day 5, and Day 10
Population: PK set. Here, the "number analyzed" signifies those participants who were evaluable for this outcome measure at specified time points.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Part B: VX-121 (Cohort B1) | Part B: VX-121 (Cohort B2) | Part B: VX-121 (Cohort B3) | Part B: VX-121 (Cohort B4)
Number analyzed (Participants) | 6 | 6 | 6 | 6
mcg/mL
  Day 1 | 0.153 (0.0260) | 0.418 (0.0667) | 0.803 (0.0529) | 1.43 (0.217)
  Day 5 | 0.497 (0.0889) | 1.41 (0.316) | 2.67 (0.564) | 4.36 (0.789)
  Day 10: number analyzed (Participants) | 6 | 6 | 5 | 5
  Day 10 | 0.574 (0.122) | 1.94 (0.410) | 3.07 (0.667) | 5.07 (0.803)

5. Secondary Outcome: Part B: Area Under the Concentration Versus Time Curve During the Dosing Interval (AUCtau) of VX-121
Time Frame: Day 1, Day 5, and Day 10
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mcg*h/mL
Arm/Group | Part B: VX-121 (Cohort B1) | Part B: VX-121 (Cohort B2) | Part B: VX-121 (Cohort B3) | Part B: VX-121 (Cohort B4)
Number analyzed (Participants) | 6 | 6 | 6 | 6
mcg*h/mL
  Day 1 | 2.62 (0.435) | 7.11 (1.27) | 14.4 (1.08) | 27.5 (4.30)
  Day 5 | 10.3 (1.84) | 30.1 (6.76) | 53.8 (10.7) | 86.6 (16.6)
  Day 10: number analyzed (Participants) | 6 | 6 | 5 | 5
  Day 10 | 11.5 (2.52) | 38.2 (9.26) | 58.7 (12.6) | 97.5 (17.2)

6. Secondary Outcome: Part B: Observed Pre-dose Plasma Concentration (Ctrough) of VX-121
Time Frame: Pre-dose at Day 5 and Day 10
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Part B: VX-121 (Cohort B1) | Part B: VX-121 (Cohort B2) | Part B: VX-121 (Cohort B3) | Part B: VX-121 (Cohort B4)
Number analyzed (Participants) | 6 | 6 | 6 | 6
mcg/mL
  Day 5 | 0.391 (0.0694) | 1.16 (0.266) | 2.07 (0.537) | 2.94 (0.759)
  Day 10: number analyzed (Participants) | 6 | 6 | 5 | 5
  Day 10 | 0.484 (0.109) | 1.64 (0.414) | 2.40 (0.637) | 3.81 (0.792)

7. Secondary Outcome: Part C: Maximum Observed Concentration (Cmax) of VX-121, TEZ and Its Metabolites (M1-TEZ and M2-TEZ) and, IVA and Its Metabolites (M1-IVA and M6-IVA)
Time Frame: Day 1, Day 7, and Day 14
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Part C: VX-121 (Cohort C1) | Part C: VX-121 (Cohort C2) | Part C: VX-121 (Cohort C3)
Number analyzed (Participants) | 6 | 7 | 6
mcg/mL
  VX-121: Day 1 | 0.212 (0.0501) | 0.408 (0.122) | 0.0728 (0.0102)
  VX-121: Day 7: number analyzed (Participants) | 5 | 6 | 6
  VX-121: Day 7 | 1.18 (0.735) | 1.77 (0.416) | 0.364 (0.122)
  VX-121: Day 14: number analyzed (Participants) | 5 | 6 | 4
  VX-121: Day 14 | 1.39 (0.651) | 2.14 (0.476) | 0.385 (0.108)
  TEZ: Day 1 | 5.97 (1.33) | 6.75 (0.936) | 5.11 (1.35)
  TEZ: Day 7: number analyzed (Participants) | 5 | 6 | 6
  TEZ: Day 7 | 9.48 (3.09) | 8.72 (0.561) | 7.50 (1.24)
  TEZ: Day 14: number analyzed (Participants) | 5 | 6 | 4
  TEZ: Day 14 | 9.49 (3.76) | 9.08 (0.547) | 7.27 (1.40)
  M1-TEZ: Day 1 | 1.09 (0.327) | 1.24 (0.399) | 1.12 (0.259)
  M1-TEZ: Day 7: number analyzed (Participants) | 5 | 6 | 6
  M1-TEZ: Day 7 | 5.07 (1.10) | 6.48 (1.48) | 5.20 (0.606)
  M1-TEZ: Day 14: number analyzed (Participants) | 5 | 6 | 4
  M1-TEZ: Day 14 | 6.44 (1.36) | 8.12 (1.41) | 6.70 (1.19)
  M2-TEZ: Day 1 | 0.521 (0.191) | 0.622 (0.390) | 0.662 (0.320)
  M2-TEZ: Day 7: number analyzed (Participants) | 5 | 6 | 6
  M2-TEZ: Day 7 | 4.79 (2.03) | 6.16 (2.17) | 5.56 (3.67)
  M2-TEZ: Day 14: number analyzed (Participants) | 5 | 6 | 4
  M2-TEZ: Day 14 | 6.45 (2.88) | 8.78 (3.54) | 9.07 (6.13)
  IVA: Day 1 | 1.02 (0.158) | 1.00 (0.235) | 0.770 (0.169)
  IVA: Day 7: number analyzed (Participants) | 5 | 6 | 6
  IVA: Day 7 | 2.15 (1.27) | 1.40 (0.288) | 1.37 (0.309)
  IVA: Day 14: number analyzed (Participants) | 5 | 6 | 4
  IVA: Day 14 | 2.14 (1.20) | 1.35 (0.231) | 1.20 (0.402)
  M1-IVA: Day 1 | 1.91 (0.573) | 2.34 (0.602) | 1.51 (0.349)
  M1-IVA: Day 7: number analyzed (Participants) | 5 | 6 | 6
  M1-IVA: Day 7 | 3.91 (1.80) | 3.42 (0.534) | 2.65 (0.434)
  M1-IVA: Day 14: number analyzed (Participants) | 5 | 6 | 4
  M1-IVA: Day 14 | 4.11 (1.86) | 2.97 (0.640) | 3.14 (1.32)
  M6-IVA: Day 1 | 0.779 (0.343) | 1.29 (0.796) | 1.24 (0.727)
  M6-IVA: Day 7: number analyzed (Participants) | 5 | 6 | 6
  M6-IVA: Day 7 | 1.52 (0.889) | 2.62 (1.20) | 1.88 (1.21)
  M6-IVA: Day 14: number analyzed (Participants) | 5 | 6 | 4
  M6-IVA: Day 14 | 1.77 (0.941) | 2.26 (0.744) | 2.55 (2.20)

8. Secondary Outcome: Part C: Area Under the Concentration Versus Time Curve During a Dosing Interval (AUCtau) of VX-121, TEZ and Its Metabolites (M1-TEZ and M2-TEZ) and IVA and Its Metabolites (M1-IVA and M6-IVA)
Time Frame: Day 1, Day 7, and Day 14
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mcg*h/mL
Arm/Group | Part C: VX-121 (Cohort C1) | Part C: VX-121 (Cohort C2) | Part C: VX-121 (Cohort C3)
Number analyzed (Participants) | 6 | 7 | 6
mcg*h/mL
  VX-121: Day 1: number analyzed (Participants) | 6 | 6 | 6
  VX-121: Day 1 | 3.51 (0.813) | 7.96 (0.789) | 1.18 (0.130)
  VX-121: Day 7: number analyzed (Participants) | 5 | 6 | 6
  VX-121: Day 7 | 21.7 (10.6) | 35.4 (8.27) | 6.52 (1.20)
  VX-121: Day 14: number analyzed (Participants) | 5 | 6 | 4
  VX-121: Day 14 | 26.6 (14.5) | 41.1 (8.29) | 7.34 (1.63)
  TEZ: Day 1 | 56.1 (16.6) | 50.9 (7.11) | 44.6 (11.5)
  TEZ: Day 7: number analyzed (Participants) | 5 | 6 | 6
  TEZ: Day 7 | 133 (51.6) | 103 (13.9) | 88.8 (21.0)
  TEZ: Day 14: number analyzed (Participants) | 5 | 6 | 4
  TEZ: Day 14 | 138 (60.8) | 112 (10.4) | 87.6 (28.6)
  M1-TEZ: Day 1 | 20.7 (7.03) | 24.9 (6.61) | 20.7 (4.99)
  M1-TEZ: Day 7: number analyzed (Participants) | 5 | 6 | 6
  M1-TEZ: Day 7 | 107 (24.8) | 130 (22.3) | 109 (14.1)
  M1-TEZ: Day 14: number analyzed (Participants) | 5 | 6 | 6
  M1-TEZ: Day 14 | 139 (29.7) | 167 (24.7) | 142 (27.0)
  M2-TEZ: Day 1 | 6.68 (2.49) | 9.61 (5.51) | 7.57 (3.18)
  M2-TEZ: Day 7: number analyzed (Participants) | 5 | 6 | 6
  M2-TEZ: Day 7 | 103 (41.1) | 130 (46.7) | 117 (72.6)
  M2-TEZ: Day 14: number analyzed (Participants) | 5 | 6 | 4
  M2-TEZ: Day 14 | 143 (64.1) | 194 (82.7) | 200 (144)
  IVA: Day 1 | 6.16 (1.36) | 5.85 (1.64) | 4.30 (0.504)
  IVA: Day 7: number analyzed (Participants) | 5 | 6 | 6
  IVA: Day 7 | 18.8 (12.3) | 11.6 (3.26) | 11.0 (3.73)
  IVA: Day 14: number analyzed (Participants) | 5 | 6 | 4
  IVA: Day 14 | 18.4 (10.7) | 11.2 (2.75) | 9.02 (2.62)
  M1-IVA: Day 1 | 11.5 (3.01) | 14.1 (1.68) | 9.37 (1.97)
  M1-IVA: Day 7: number analyzed (Participants) | 5 | 6 | 6
  M1-IVA: Day 7 | 32.6 (17.3) | 27.3 (4.79) | 22.3 (3.70)
  M1-IVA: Day 14: number analyzed (Participants) | 5 | 6 | 4
  M1-IVA: Day 14 | 32.2 (17.3) | 25.3 (4.35) | 24.2 (12.3)
  M6-IVA: Day 1 | 4.08 (1.63) | 9.42 (4.83) | 4.99 (2.99)
  M6-IVA: Day 7: number analyzed (Participants) | 5 | 6 | 6
  M6-IVA: Day 7 | 15.2 (9.34) | 26.5 (12.7) | 19.2 (12.8)
  M6-IVA: Day 14: number analyzed (Participants) | 5 | 6 | 4
  M6-IVA: Day 14 | 17.6 (10.2) | 22.6 (8.19) | 26.4 (24.3)

9. Secondary Outcome: Part C: Pre-dose Plasma Concentration (Ctrough) of VX-121, TEZ and Its Metabolites (M1-TEZ and M2-TEZ) and IVA and Its Metabolites (M1-IVA and M6-IVA)
Time Frame: Pre-dose at Day 7 and Day 14
Population: PK set. Here, the "overall number of participants analyzed" signifies those participants who were evaluable for this outcome measure and "number analyzed" signifies those participants who were evaluable for this outcome measure at specified timepoints.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Part C: VX-121 (Cohort C1) | Part C: VX-121 (Cohort C2) | Part C: VX-121 (Cohort C3)
Number analyzed (Participants) | 5 | 6 | 6
mcg/mL
  VX-121: Day 7 | 0.916 (0.369) | 1.37 (0.321) | 0.258 (0.0426)
  VX-121: Day 14: number analyzed (Participants) | 5 | 6 | 4
  VX-121: Day 14 | 1.24 (0.665) | 1.72 (0.452) | 0.357 (0.0966)
  TEZ: Day 7 | 3.95 (1.84) | 2.57 (0.776) | 2.31 (0.735)
  TEZ: Day 14: number analyzed (Participants) | 5 | 6 | 4
  TEZ: Day 14 | 4.55 (2.50) | 3.27 (0.646) | 2.27 (0.851)
  M1-TEZ: Day 7 | 4.09 (1.22) | 4.53 (0.512) | 3.96 (0.685)
  M1-TEZ: Day 14: number analyzed (Participants) | 5 | 6 | 4
  M1-TEZ: Day 14 | 5.45 (1.46) | 6.40 (1.17) | 5.03 (1.18)
  M2-TEZ: Day 7 | 4.30 (1.66) | 5.08 (2.06) | 4.75 (2.97)
  M2-TEZ: Day 14: number analyzed (Participants) | 5 | 6 | 4
  M2-TEZ: Day 14 | 6.20 (2.60) | 5.51 (1.72) | 8.63 (6.24)
  IVA: Day 7 | 1.33 (0.834) | 0.768 (0.230) | 0.780 (0.317)
  IVA: Day 14: number analyzed (Participants) | 5 | 6 | 4
  IVA: Day 14 | 1.34 (0.889) | 0.750 (0.252) | 0.601 (0.164)
  M1-IVA: Day 7 | 2.46 (1.53) | 2.00 (0.589) | 1.67 (0.334)
  M1-IVA: Day 14: number analyzed (Participants) | 5 | 6 | 4
  M1-IVA: Day 14 | 2.45 (1.37) | 1.87 (0.509) | 1.73 (0.977)
  M6-IVA: Day 7 | 1.28 (0.763) | 2.09 (1.11) | 1.67 (1.31)
  M6-IVA: Day 14: number analyzed (Participants) | 5 | 6 | 4
  M6-IVA: Day 14 | 1.60 (0.926) | 1.85 (0.738) | 2.27 (2.26)

10. Secondary Outcome: Part D: Maximum Observed Concentration (Cmax) of VX-121, TEZ and Its Metabolites (M1-TEZ and M2-TEZ) and IVA and Its Metabolites (M1-IVA and M6-IVA)
Time Frame: Day 1 and Day 15
Population: PK set.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Part D: VX-121/TEZ/IVA
Number analyzed (Participants) | 9
mcg/mL
  VX-121: Day 1 | 0.0553 (0.0207)
  VX-121: Day 15 | 0.389 (0.116)
  TEZ: Day 1 | 5.38 (1.39)
  TEZ: Day 15 | 6.80 (2.13)
  M1-TEZ: Day 1 | 1.26 (0.162)
  M1-TEZ: Day 15 | 5.56 (1.19)
  M2-TEZ: Day 1 | 0.243 (0.0629)
  M2-TEZ: Day 15 | 3.99 (1.41)
  IVA: Day 1 | 0.745 (0.279)
  IVA: Day 15 | 1.47 (0.472)
  M1-IVA: Day 1 | 1.34 (0.478)
  M1-IVA: Day 15 | 2.69 (0.829)
  M6-IVA: Day 1 | 0.531 (0.229)
  M6-IVA: Day 15 | 1.17 (0.589)

11. Secondary Outcome: Part D: Area Under the Concentration Versus Time Curve From the Time of Dosing to the Last Measurable Concentration (AUC[0-last]) of VX-121, TEZ and Its Metabolites (M1-TEZ and M2-TEZ) and IVA and Its Metabolites (M1-IVA and M6-IVA)
Time Frame: Day 1 and Day 15
Population: PK set.
Measure: Mean (Standard Deviation); unit: mcg*h/mL
Arm/Group | Part D: VX-121/TEZ/IVA
Number analyzed (Participants) | 9
mcg*h/mL
  VX-121: Day 1 | 0.160 (0.0766)
  VX-121: Day 15 | 2.50 (1.07)
  TEZ: Day 1 | 21.9 (5.48)
  TEZ: Day 15 | 37.4 (16.0)
  M1-TEZ: Day 1 | 4.66 (1.42)
  M1-TEZ: Day 15 | 37.8 (14.3)
  M2-TEZ: Day 1 | 0.630 (0.213)
  M2-TEZ: Day 15 | 28.6 (13.7)
  IVA: Day 1 | 2.74 (1.24)
  IVA: Day 15 | 9.27 (4.06)
  M1-IVA: Day 1 | 4.51 (1.97)
  M1-IVA: Day 15 | 16.4 (6.70)
  M6-IVA: Day 1 | 1.25 (0.529)
  M6-IVA: Day 15 | 7.58 (4.49)

12. Secondary Outcome: Part D: Pre-dose Plasma Concentration (Ctrough) of VX-121, TEZ and Its Metabolites (M1-TEZ and M2-TEZ) and IVA and Its Metabolites (M1-IVA and M6-IVA)
Time Frame: Pre-dose at Day 8, Day 15, and Day 29
Population: PK set.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Part D: VX-121/TEZ/IVA
Number analyzed (Participants) | 9
mcg/mL
  VX-121: Day 8 | 0.258 (0.0834)
  VX-121: Day 15 | 0.348 (0.109)
  VX-121: Day 29 | 0.323 (0.110)
  TEZ: Day 8 | 1.78 (0.525)
  TEZ: Day 15 | 2.01 (0.543)
  TEZ: Day 29 | 2.02 (0.927)
  M1-TEZ: Day 8 | 4.15 (0.648)
  M1-TEZ: Day 15 | 4.52 (1.06)
  M1-TEZ: Day 29 | 5.11 (1.50)
  M2-TEZ: Day 8 | 3.29 (1.41)
  M2-TEZ: Day 15 | 3.76 (1.29)
  M2-TEZ: Day 29 | 4.57 (2.28)
  IVA: Day 8 | 0.873 (0.367)
  IVA: Day 15 | 0.998 (0.367)
  IVA: Day 29 | 0.916 (0.586)
  M1-IVA: Day 8 | 1.38 (0.427)
  M1-IVA: Day 15 | 1.76 (0.619)
  M1-IVA: Day 29 | 1.62 (0.620)
  M6-IVA: Day 8 | 0.823 (0.573)
  M6-IVA: Day 15 | 0.819 (0.412)
  M6-IVA: Day 29 | 0.990 (0.632)

13. Secondary Outcome: Part D: Absolute Change in Sweat Chloride (SwCl) Concentrations
Description: Sweat samples were collected using an approved collection device.
Time Frame: From Baseline Through Day 29
Population: Full analysis set (FAS) included all randomized participants who carry the intended CF transmembrane conductance regulator protein (CFTR) allele mutation and have received at least 1 dose of study drug in the treatment period.
Measure: Least Squares Mean (95% Confidence Interval); unit: millimole per liter (mmol/L)
Arm/Group | Part D: Placebo | Part D: VX-121/TEZ/IVA
Number analyzed (Participants) | 3 | 9
millimole per liter (mmol/L) | 2.6 [-19.7 to 24.9] | -47.7 [-58.2 to -37.2]

14. Secondary Outcome: Part D: Absolute Change in Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1)
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration.
Time Frame: From Baseline Through Day 29
Population: FAS.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage points
Arm/Group | Part D: Placebo | Part D: VX-121/TEZ/IVA
Number analyzed (Participants) | 3 | 9
percentage points | -2.0 [-12.9 to 8.9] | 8.3 [2.8 to 13.8]

ADVERSE EVENTS:
Time Frame: From Day 1 Through Safety Follow-up (up to Day 15 for Part A [except Cohorts A3 and A9], up to Day 26 for Cohort A3, up to Day 34 for Cohort A9, up to Day 20 for Part B, up to Day 24 for Part C and up to Week 9 for Part D)
Arm/Group | Part A: Pooled Placebo (Cohorts A1-5; Except A3) | Part A: VX-121 (Cohort A1) | Part A: VX-121 (Cohort A2) | Part A: VX-121 (Cohort A3) | Part A: VX-121 (Cohort A4) | Part A: VX-121 (Cohort A5) | Part A: VX-121 (Cohort A9) | Part B: Pooled Placebo (Cohorts B1-4) | Part B: VX-121 (Cohort B1) | Part B: VX-121 (Cohort B2) | Part B: VX-121 (Cohort B3) | Part B: VX-121 (Cohort B4) | Part C: Pooled Placebo (Cohorts C1-3) | Part C: VX-121 (Cohort C1) | Part C: VX-121 (Cohort C2) | Part C: VX-121 (Cohort C3) | Part D: Placebo | Part D: VX-121/TEZ/IVA
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/5 | 0/6 | 0/6 | 0/6 | 0/6 | 0/8 | 0/9 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/7 | 0/6 | 0/3 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/5 | 0/6 | 0/6 | 0/6 | 0/6 | 0/8 | 0/9 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/7 | 0/6 | 1/3 | 0/9
Other Adverse Events (participants affected / at risk) | 1/8 | 4/5 | 2/6 | 4/6 | 1/6 | 2/6 | 7/8 | 7/9 | 3/6 | 5/6 | 4/6 | 5/6 | 4/6 | 3/6 | 6/7 | 3/6 | 2/3 | 7/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Pooled Placebo (Cohorts A1-5; Except A3) (N=8) | Part A: VX-121 (Cohort A1) (N=5) | Part A: VX-121 (Cohort A2) (N=6) | Part A: VX-121 (Cohort A3) (N=6) | Part A: VX-121 (Cohort A4) (N=6) | Part A: VX-121 (Cohort A5) (N=6) | Part A: VX-121 (Cohort A9) (N=8) | Part B: Pooled Placebo (Cohorts B1-4) (N=9) | Part B: VX-121 (Cohort B1) (N=6) | Part B: VX-121 (Cohort B2) (N=6) | Part B: VX-121 (Cohort B3) (N=6) | Part B: VX-121 (Cohort B4) (N=6) | Part C: Pooled Placebo (Cohorts C1-3) (N=6) | Part C: VX-121 (Cohort C1) (N=6) | Part C: VX-121 (Cohort C2) (N=7) | Part C: VX-121 (Cohort C3) (N=6) | Part D: Placebo (N=3) | Part D: VX-121/TEZ/IVA (N=9)
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Pooled Placebo (Cohorts A1-5; Except A3) (N=8) | Part A: VX-121 (Cohort A1) (N=5) | Part A: VX-121 (Cohort A2) (N=6) | Part A: VX-121 (Cohort A3) (N=6) | Part A: VX-121 (Cohort A4) (N=6) | Part A: VX-121 (Cohort A5) (N=6) | Part A: VX-121 (Cohort A9) (N=8) | Part B: Pooled Placebo (Cohorts B1-4) (N=9) | Part B: VX-121 (Cohort B1) (N=6) | Part B: VX-121 (Cohort B2) (N=6) | Part B: VX-121 (Cohort B3) (N=6) | Part B: VX-121 (Cohort B4) (N=6) | Part C: Pooled Placebo (Cohorts C1-3) (N=6) | Part C: VX-121 (Cohort C1) (N=6) | Part C: VX-121 (Cohort C2) (N=7) | Part C: VX-121 (Cohort C3) (N=6) | Part D: Placebo (N=3) | Part D: VX-121/TEZ/IVA (N=9)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eye irritation (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Defaecation urgency (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site bruise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0
Catheter site erythema (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site irritation (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site pain (General disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Catheter site pruritus (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Feeling cold (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Feeling hot (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Injection site bruising (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Puncture site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vessel puncture site bruise (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vessel puncture site pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0
Periodontitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Faecal volume decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Influenza A virus test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 2 | 2 | 0 | 0 | 0
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 2 | 1 | 0 | 0 | 4 | 2 | 2 | 0 | 0 | 1 | 1 | 0 | 4 | 2 | 0 | 1
Nerve compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ophthalmoplegic migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tension (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Papule (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin hypertrophy (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-07-27): https://cdn.clinicaltrials.gov/large-docs/89/NCT03768089/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-28): https://cdn.clinicaltrials.gov/large-docs/89/NCT03768089/SAP_001.pdf